CLINICAL TRIAL: NCT01144377
Title: A Phase 2 Randomized Study of LY2541546 Versus Placebo in Postmenopausal Women With Low Bone Mineral Density: An Evaluation of the Dose Response Relationship Using Bone Mineral Density
Brief Title: A Study of LY2541546 in Women With Low Bone Mineral Density
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11953; I2M-MC-GSDB (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-06-11; First posted 2010-06-15 (Estimated); Results first posted 2017-12-04 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Osteoporosis
Keywords: osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — blosozumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 180 mg LY2541546 Q4W + Placebo (Experimental): LY2541546: 180 milligrams (mg) administered subcutaneously every 4 weeks (Q4W) for 52 weeks.
  Placebo: administered subcutaneously every alternate 2 weeks from the LY2541546 dose for 52 weeks.
  Interventions: Drug: LY2541546; Drug: Placebo
- 180 mg LY2541546 Q2W (Experimental): LY2541546: 180 milligrams (mg) administered subcutaneously every 2 weeks (Q2W) for 52 weeks.
  Interventions: Drug: LY2541546
- 270 mg LY2541546 Q2W (Experimental): LY2541546: 270 milligrams (mg) LY2541546 administered subcutaneously every 2 weeks (Q2W) for 52 weeks.
  Interventions: Drug: LY2541546
- 270 mg LY2541546 Q12W + Placebo (Experimental): LY2541546: 270 milligrams (mg) administered subcutaneously every 12 weeks (Q12W) for 52 weeks.
  Placebo: administered subcutaneously every alternate 2 weeks from the LY2541546 dose for 52 weeks.
  Interventions: Drug: LY2541546; Drug: Placebo
- Placebo Comparator Q2W (Placebo Comparator): Placebo: administered subcutaneously every 2 weeks (Q2W) for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2541546 — Administered subcutaneously
  Other Names: Blosozumab
  Arms: 180 mg LY2541546 Q2W; 180 mg LY2541546 Q4W + Placebo; 270 mg LY2541546 Q12W + Placebo; 270 mg LY2541546 Q2W
Drug: Placebo — Administered subcutaneously
  Arms: 180 mg LY2541546 Q4W + Placebo; 270 mg LY2541546 Q12W + Placebo; Placebo Comparator Q2W

SUMMARY:
The primary objectives of this study include evaluating the dose response of LY2541546 using bone mineral density (BMD) change from baseline as compared to placebo and evaluating the overall safety and tolerability of LY2541546 following multiple subcutaneous administrations in postmenopausal (PMP) women with low BMD. Following the last dose of study drug, participants will be able to participate in a 12 month extension to collect additional safety and efficacy data (no further treatment will be administered during this extension).

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory, postmenopausal women, inclusive.
* Have low bone mineral density (BMD), defined as a T-score or equivalent BMD absolute value (grams/square centimeter [g/cm^2]) for the lumbar spine of between -3.5 and -2.0, inclusive.
* Without language barrier, reliable, and willing to make themselves available for the duration of the study and to follow study procedures.
* Willing to take study drug and daily supplements (calcium and Vitamin D).
* Normal laboratory tests or laboratory test results determined not clinically significant by the investigator. Serum phosphate and serum calcium must be within normal limits, and platelet level greater than 100,000 cubic millimeters (mm^3).

Exclusion Criteria:

* Have received treatment with any of the following medications more recently than 3 months prior to screening Androgen, Calcitonin, Estrogen (including over the counter preparations known to have estrogenic activity), Progestin (including over the counter preparations known to have progestogenic activity), selective estrogen receptor modulators (SERMs) (Raloxifene, Tamoxifen, Toremifene, Clomiphene), or Tibolone.
* Have previously used or currently use denosumab, parathyroid hormone (PTH) and/or PTH analogs, strontium ranelate, or parenteral formulations of bisphosphonates.
* Have received treatment with any oral bisphosphonate within the last year.
* Have received therapeutic doses of systemic corticosteroids for more than one month during the 6 months prior to screening.
* Have received therapeutic doses of fluorides (20 milligrams per day) for more than 3 months during the last 3 years, or for more than a total of 2 years, or any within the last 6 months.
* Have severe Vitamin D deficiency defined as 25-hydroxyvitamin D less than <9.2 nanograms per milliliter (ng/mL) [23 nanomoles per liter (nmol/L)] at screening. If the serum 25-hydroxy-vitamin D level at screening is less than or equal to 9.2 ng/mL and <20 ng/mL, participants will receive a loading dose of Vitamin D (at a dose of approximately 100,000 international units (IU) given orally) prior to enrollment.
* Have any known bone disorder other than low BMD or osteoporosis.
* Have a history of osteoporotic fractures, including known prevalent vertebral fracture or evidence of prevalent vertebral fracture on screening spine X-ray or dual-energy x-ray absorptiometry (DXA), or are considered to be at high risk for fracture.
* Presence of any abnormality (such as artifacts or osteophytes) that would confound DXA evaluation of lumbar vertebrae in the L-1 through L-4 region.
* Have a history of Bell's palsy, other cranial nerve disorders, or have a history of Temporomandibular Joint and Muscle Disorders (TMJDs).
* Have any history of cancer within the previous 5 years, except for excised superficial lesions such as basal cell carcinoma and squamous cell carcinoma of the skin.
* Have history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of constituting a risk when taking the study medication or of interfering with the interpretation of data.
* Have acute or chronic liver disease ([bilirubin >34 micromoles per liter (µmol/L) or >2.0 milligrams per deciliter (mg/dL), alanine transaminase [ALT/SGPT] >100 units per liter (U/L), or alkaline phosphatase >300 U/L)].
* Have impaired kidney function serum creatinine >135 µmol/L or >2.0 mg/dL.
* Have known allergy to LY2541546, any of diluents or excipients of LY2541546, or significant allergy to any other monoclonal antibody.
* History of excessive consumption of alcohol or abuse of drugs within the last year.
* Have poor medical condition or psychiatric risks for treatment with an investigational drug.

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2010-08; Primary Completion 2012-05 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (8):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bethesda, Maryland
- Denmark (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hvidovre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vejle
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tallinn, Estonia
- Japan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After exposure to study medication for the 52 week treatment phase, participants entered a 12 week non-treatment safety follow-up period with the option of staying in the non-treatment safety follow-up period for an additional 40 weeks (for a total of 52 weeks follow-up for the main study participants only).
Groups:
- 180 mg LY2541546 Q4W + Placebo: LY2541546 + Placebo: 180 milligrams (mg) LY2541546 administered subcutaneously every 4 weeks (Q4W) for 52 weeks with Placebo administered subcutaneously every alternate 2 weeks from the LY2541546 dose for 52 weeks. After exposure to study medication for the 52 week treatment phase, participants entered a 12 week non-treatment safety follow-up period with the option of staying in the non-treatment safety follow-up period for an additional 40 weeks (for a total of 52 weeks follow-up for the main study participants only).
- 180 mg LY2541546 Q2W: LY2541546: 180 mg administered subcutaneously every 2 weeks (Q2W) for 52 weeks. After exposure to study medication for the 52 week treatment phase, participants entered a 12 week non-treatment safety follow-up period with the option of staying in the non-treatment safety follow-up period for an additional 40 weeks (for a total of 52 weeks follow-up for the main study participants only).
- 270 mg LY2541546 Q2W: LY2541546: 270 mg administered subcutaneously every 2 weeks (Q2W) for 52 weeks. After exposure to study medication for the 52 week treatment phase, participants entered a 12 week non-treatment safety follow-up period with the option of staying in the non-treatment safety follow-up period for an additional 40 weeks (for a total of 52 weeks follow-up for the main study participants only).
- 270 mg LY2541546 Q12W + Placebo: LY2541546 + Placebo: 270 mg LY2541546 administered subcutaneously every 12 weeks (Q12W) with Placebo administered subcutaneously every 2 weeks when LY2541546 is not administered for 52 weeks. After exposure to study medication for the 52 week treatment phase, participants entered a 12 week non-treatment safety follow-up period with the option of staying in the non-treatment safety follow-up period for an additional 40 weeks (for a total of 52 weeks follow-up for the main study participants only).
- Placebo Q2W: Placebo: administered subcutaneously every 2 weeks (Q2W) for 52 weeks. After exposure to study medication for the 52 week treatment phase, participants entered a 12 week non-treatment safety follow-up period with the option of staying in the non-treatment safety follow-up period (for an additional 40 weeks for a total of 52 weeks follow-up for the main study participants only).
Period: 52 Week Treatment Period
Arm/Group | 180 mg LY2541546 Q4W + Placebo | 180 mg LY2541546 Q2W | 270 mg LY2541546 Q2W | 270 mg LY2541546 Q12W + Placebo | Placebo Q2W
Started | 31 | 30 | 30 | 26 | 37
Received at Least One Dose of Study Drug | 31 | 30 | 30 | 25 | 37
Completed | 26 | 29 | 25 | 22 | 34
Not Completed | 5 | 1 | 5 | 4 | 3
Not completed — Adverse Event | 0 | 0 | 3 | 2 | 1
Not completed — Entry Criteria Not Met | 0 | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 1 | 1 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 1
Period: 12 Week Safety Follow-up Period
Arm/Group | 180 mg LY2541546 Q4W + Placebo | 180 mg LY2541546 Q2W | 270 mg LY2541546 Q2W | 270 mg LY2541546 Q12W + Placebo | Placebo Q2W
Started | 26 | 29 | 25 | 22 | 34
Completed | 26 (Of the 26 participants who completed this Period, 22 continued to the Optional 40 Week follow-up.) | 29 (Of the 29 participants who completed this Period, 25 continued to the Optional 40 Week follow-up.) | 25 (Of the 25 participants who completed this Period, 23 continued to the Optional 40 Week follow-up.) | 22 (Of the 22 participants who completed this Period, 3 continued to the Optional 40 Week follow-up.) | 34 (Of the 34 participants who completed this Period, 23 continued to the Optional 40 Week follow-up.)
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Optional 40 Week Safety Follow-up Period
Arm/Group | 180 mg LY2541546 Q4W + Placebo | 180 mg LY2541546 Q2W | 270 mg LY2541546 Q2W | 270 mg LY2541546 Q12W + Placebo | Placebo Q2W
Started | 22 | 25 | 23 | 3 | 23
Completed | 21 | 24 | 23 | 3 | 21
Not Completed | 1 | 1 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Sponsor Decision | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of study drug.
Groups:
- 180 mg LY2541546 Q4W + Placebo: LY2541546 + Placebo: 180 milligrams (mg) LY2541546 administered subcutaneously every 4 weeks (Q4W) for 52 weeks with Placebo administered subcutaneously every alternate 2 weeks from the LY2541546 dose for 52 weeks.
- 180 mg LY2541546 Q2W: LY2541546: 180 mg administered subcutaneously every 2 weeks (Q2W) for 52 weeks.
- 270 mg LY2541546 Q2W: LY2541546: 270 mg administered subcutaneously every 2 weeks (Q2W) for 52 weeks.
- 270 mg LY2541546 Q12W + Placebo: LY2541546 + Placebo: 270 mg LY2541546 administered subcutaneously every 12 weeks (Q12W) with Placebo administered subcutaneously every 2 weeks when LY2541546 is not administered for 52 weeks.
- Placebo Q2W: Placebo: administered subcutaneously every 2 weeks (Q2W) for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | 180 mg LY2541546 Q4W + Placebo | 180 mg LY2541546 Q2W | 270 mg LY2541546 Q2W | 270 mg LY2541546 Q12W + Placebo | Placebo Q2W | Total
Number analyzed (Participants) | 31 | 30 | 30 | 25 | 37 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.78 (8.98) | 64.17 (8.20) | 66.12 (7.68) | 63.56 (8.02) | 65.17 (8.91) | 65.22 (8.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 30 | 25 | 37 | 153
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 2 | 9 | 8 | 27
  Not Hispanic or Latino | 23 | 24 | 26 | 16 | 26 | 115
  Unknown or Not Reported | 4 | 2 | 2 | 0 | 3 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 14 | 13 | 13 | 11 | 14 | 65
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1
  White | 17 | 17 | 17 | 14 | 22 | 87
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 6 | 5 | 11 | 10 | 36
  Estonia | 4 | 3 | 5 | 3 | 4 | 19
  Lithuania | 3 | 4 | 4 | 0 | 4 | 15
  Denmark | 6 | 4 | 3 | 0 | 5 | 18
  Japan | 14 | 13 | 13 | 11 | 14 | 65
Lumbar Spine Bone Mineral Density (Baseline) [Mean (Standard Deviation); unit: grams/square centimeter (g/cm^2)] | 0.78 (0.09) | 0.78 (0.07) | 0.80 (0.09) | 0.77 (0.09) | 0.78 (0.09) | 0.78 (0.09)
Femoral Neck Bone Mineral Density (Baseline) [Mean (Standard Deviation); unit: g/cm^2] | 0.66 (0.15) | 0.66 (0.15) | 0.69 (0.11) | 0.63 (0.11) | 0.66 (0.17) | 0.66 (0.14)
Total Hip Bone Mineral Density (Baseline) [Mean (Standard Deviation); unit: grams/square centimeter] | 0.75 (0.11) | 0.75 (0.13) | 0.77 (0.10) | 0.73 (0.11) | 0.73 (0.14) | 0.75 (0.12)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 52 Week Endpoint in Lumbar Spine Bone Mineral Density (BMD)
Description: Lumbar spine bone mineral density (BMD) measured by dual energy x-ray absorptiometry (DXA).
  Least squares (LS) mean values were determined using a mixed-effects model repeated-measures (MMRM) analysis of covariance.
  Factors in the model included treatment, time and the interaction of treatment by time as fixed effects, and baseline lumbar spine BMD as a covariate.
Time Frame: Baseline, 52 weeks
Population: Participants who received at least one dose of study drug with baseline and at least one post-baseline lumbar spine BMD value.
Measure: Least Squares Mean (95% Confidence Interval); unit: g/cm^2
Groups:
- 180 mg LY2541546 Q4W + Placebo: LY2541546 + Placebo: 180 milligrams (mg) LY2541546 administered subcutaneously every 4 weeks (Q4W) for 52 weeks with Placebo administered every alternate 2 weeks from the LY2541546 dose for 52 weeks.
- 270 mg LY2541546 Q12W + Placebo: LY2541546 + Placebo: 270 mg LY2541546 administered subcutaneously every 12 weeks (Q12W) with Placebo administered every 2 weeks when LY2541546 is not administered for 52 weeks.
Arm/Group | 180 mg LY2541546 Q4W + Placebo | 180 mg LY2541546 Q2W | 270 mg LY2541546 Q2W | 270 mg LY2541546 Q12W + Placebo | Placebo Q2W
Number analyzed (Participants) | 27 | 29 | 26 | 22 | 34
g/cm^2 | 0.065 [0.048 to 0.082] | 0.115 [0.099 to 0.131] | 0.142 [0.125 to 0.158] | 0.054 [0.036 to 0.073] | -0.011 [-0.026 to 0.004]

2. Secondary Outcome: Change From Baseline to 12, 24, and 64 Weeks in Lumbar Spine Bone Mineral Density (BMD)
Description: as for outcome 1
Time Frame: Baseline, 12 weeks and 24 weeks and 64 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: g/cm^2
Arm/Group | 180 mg LY2541546 Q4W + Placebo | 180 mg LY2541546 Q2W | 270 mg LY2541546 Q2W | 270 mg LY2541546 Q12W + Placebo | Placebo Q2W
Number analyzed (Participants) | 29 | 30 | 30 | 24 | 36
g/cm^2
  Week 12: number analyzed (Participants) | 29 | 30 | 29 | 24 | 35
  Week 12 | 0.028 [0.020 to 0.037] | 0.048 [0.039 to 0.057] | 0.057 [0.048 to 0.065] | 0.039 [0.029 to 0.049] | -0.007 [-0.015 to 0.001]
  Week 24: number analyzed (Participants) | 27 | 29 | 28 | 23 | 36
  Week 24 | 0.049 [0.037 to 0.061] | 0.083 [0.071 to 0.094] | 0.098 [0.086 to 0.109] | 0.048 [0.035 to 0.061] | -0.006 [-0.016 to 0.004]
  Week 64: number analyzed (Participants) | 26 | 29 | 25 | 22 | 34
  Week 64 | 0.046 [0.032 to 0.061] | 0.098 [0.083 to 0.112] | 0.135 [0.120 to 0.150] | 0.046 [0.029 to 0.062] | -0.007 [-0.020 to 0.006]

3. Secondary Outcome: Change From Baseline to 24, 52, and 64 Weeks in Proximal Femur Bone Mineral Density (BMD)
Description: Femoral neck and total hip bone mineral density (BMD) measured by dual energy x-ray absorptiometry (DXA).
  Least squares (LS) mean values were determined using a mixed-effects model repeated-measures (MMRM) analysis of covariance.
  Factors in the model included treatment, time and the interaction of treatment by time as fixed effects, and baseline BMD as a covariate.
Time Frame: Baseline, 24 weeks and 52 weeks and 64 weeks
Population: Participants who received at least one dose of study drug with baseline and at least one post-baseline femoral neck or total hip BMD value.
Measure: Least Squares Mean (95% Confidence Interval); unit: g/cm^2
Arm/Group | 180 mg LY2541546 Q4W + Placebo | 180 mg LY2541546 Q2W | 270 mg LY2541546 Q2W | 270 mg LY2541546 Q12W + Placebo | Placebo Q2W
Number analyzed (Participants) | 27 | 29 | 28 | 23 | 36
g/cm^2
  Femoral Neck BMD Week 24: number analyzed (Participants) | 25 | 28 | 27 | 22 | 35
  Femoral Neck BMD Week 24 | 0.010 [0.002 to 0.019] | 0.017 [0.009 to 0.025] | 0.026 [0.018 to 0.034] | 0.002 [-0.007 to 0.011] | 0.002 [-0.005 to 0.009]
  Total Hip BMD Week 24: number analyzed (Participants) | 25 | 28 | 27 | 22 | 35
  Total Hip BMD Week 24 | 0.007 [-0.001 to 0.014] | 0.020 [0.013 to 0.027] | 0.031 [0.024 to 0.039] | 0.015 [0.007 to 0.023] | -0.007 [-0.014 to -0.001]
  Femoral Neck BMD Week 52: number analyzed (Participants) | 27 | 29 | 26 | 22 | 34
  Femoral Neck BMD Week 52 | 0.018 [0.010 to 0.026] | 0.025 [0.017 to 0.033] | 0.044 [0.035 to 0.052] | 0.014 [0.005 to 0.024] | 0.003 [-0.005 to 0.010]
  Total Hip BMD Week 52: number analyzed (Participants) | 27 | 29 | 26 | 22 | 34
  Total Hip BMD Week 52 | 0.017 [0.008 to 0.025] | 0.032 [0.023 to 0.040] | 0.051 [0.043 to 0.060] | 0.019 [0.009 to 0.029] | -0.004 [-0.012 to 0.003]
  Femoral Neck BMD Week 64: number analyzed (Participants) | 26 | 29 | 25 | 22 | 34
  Femoral Neck BMD Week 64 | 0.016 [0.007 to 0.026] | 0.028 [0.019 to 0.037] | 0.038 [0.029 to 0.048] | 0.013 [0.002 to 0.023] | 0.002 [-0.007 to 0.010]
  Total Hip BMD Week 64: number analyzed (Participants) | 26 | 29 | 25 | 22 | 34
  Total Hip BMD Week 64 | 0.011 [0.001 to 0.020] | 0.031 [0.022 to 0.040] | 0.047 [0.038 to 0.056] | 0.021 [0.011 to 0.030] | -0.007 [-0.015 to 0.001]

4. Secondary Outcome: Change From Baseline to 52 Week Endpoint in Wrist Bone Mineral Density (BMD)
Description: Total radius of the wrist bone mineral density (BMD) measured by dual energy x-ray absorptiometry (DXA).
  Least squares (LS) mean values were determined using a 1-factor analysis of covariance model with treatment group as the main effect and baseline BMD as a covariate.
Time Frame: Baseline, 52 weeks
Population: Participants who received at least one dose of study drug with baseline and at least one post-baseline total radius of the wrist BMD value.
Measure: Least Squares Mean (95% Confidence Interval); unit: g/cm^2
Arm/Group | 180 mg LY2541546 Q4W + Placebo | 180 mg LY2541546 Q2W | 270 mg LY2541546 Q2W | 270 mg LY2541546 Q12W + Placebo | Placebo Q2W
Number analyzed (Participants) | 24 | 29 | 26 | 22 | 32
g/cm^2 | -0.005 [-0.011 to 0.001] | -0.005 [-0.010 to 0.001] | -0.001 [-0.007 to 0.005] | -0.002 [-0.009 to 0.004] | -0.005 [-0.010 to 0.000]

5. Secondary Outcome: Change From Baseline to 52 Week Endpoint in Bone-specific Alkaline Phosphatase (BSAP)
Time Frame: Baseline, 52 weeks
Population: Participants who received at least one dose of study drug with baseline and at least one post-baseline bone-specific alkaline phosphatase value.
Measure: Median (Inter-Quartile Range); unit: units/liter
Arm/Group | 180 mg LY2541546 Q4W + Placebo | 180 mg LY2541546 Q2W | 270 mg LY2541546 Q2W | 270 mg LY2541546 Q12W + Placebo | Placebo Q2W
Number analyzed (Participants) | 27 | 29 | 26 | 22 | 33
units/liter | -6.000 [-12.600 to 0.300] | -2.000 [-10.400 to 4.500] | 1.600 [-4.400 to 9.800] | -3.150 [-10.000 to 2.900] | -3.900 [-11.400 to 4.300]

6. Secondary Outcome: Change From Baseline to 52 Week Endpoint in Serum Type I Collagen Fragment (CTx)
Time Frame: Baseline, 52 weeks
Population: Participants who received at least one dose of study drug with baseline and at least one post-baseline serum type I collagen fragment value.
Measure: Median (Inter-Quartile Range); unit: nanograms/milliliter
Arm/Group | 180 mg LY2541546 Q4W + Placebo | 180 mg LY2541546 Q2W | 270 mg LY2541546 Q2W | 270 mg LY2541546 Q12W + Placebo | Placebo Q2W
Number analyzed (Participants) | 26 | 29 | 25 | 21 | 32
nanograms/milliliter | -0.014 [-0.116 to 0.079] | -0.088 [-0.191 to 0.030] | -0.038 [-0.199 to -0.009] | -0.022 [-0.076 to 0.029] | 0.037 [-0.076 to 0.129]

7. Secondary Outcome: Change From Baseline to 52 Week Endpoint in Osteocalcin
Time Frame: Baseline, 52 weeks
Population: Participants who received at least one dose of study drug with baseline and at least one post-baseline osteocalcin value.
Measure: Median (Inter-Quartile Range); unit: micrograms/liter
Arm/Group | 180 mg LY2541546 Q4W + Placebo | 180 mg LY2541546 Q2W | 270 mg LY2541546 Q2W | 270 mg LY2541546 Q12W + Placebo | Placebo Q2W
Number analyzed (Participants) | 26 | 29 | 25 | 22 | 32
micrograms/liter | -2.087 [-3.998 to 2.411] | -0.764 [-7.762 to 3.704] | 0.823 [-3.704 to 5.116] | -3.322 [-5.586 to 4.822] | -2.029 [-6.880 to 2.587]

8. Secondary Outcome: Change From Baseline to 52 Week Endpoint in Serum N-terminal Extension Propeptide of Type I Collagen (P1NP)
Time Frame: Baseline, 52 weeks
Population: Participants who received at least one dose of study drug with baseline and at least one post-baseline serum N-terminal extension propeptide of type I collagen value.
Measure: Median (Inter-Quartile Range); unit: nanograms/milliliter
Arm/Group | 180 mg LY2541546 Q4W + Placebo | 180 mg LY2541546 Q2W | 270 mg LY2541546 Q2W | 270 mg LY2541546 Q12W + Placebo | Placebo Q2W
Number analyzed (Participants) | 26 | 29 | 25 | 22 | 32
nanograms/milliliter | -12.250 [-19.300 to 1.300] | -4.200 [-27.200 to 6.700] | -1.100 [-12.800 to 10.200] | -16.050 [-21.700 to 0.100] | -5.800 [-11.550 to 5.450]

ADVERSE EVENTS:
Arm/Group | 180 mg LY2541546 Q4W + Placebo | 180 mg LY2541546 Q2W | 270 mg LY2541546 Q2W | 270 mg LY2541546 Q12W + Placebo | Placebo Q2W
Serious Adverse Events (participants affected / at risk) | 4/31 | 3/30 | 4/30 | 1/25 | 2/37
Other Adverse Events (participants affected / at risk) | 30/31 | 28/30 | 29/30 | 21/25 | 34/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 180 mg LY2541546 Q4W + Placebo (N=31) | 180 mg LY2541546 Q2W (N=30) | 270 mg LY2541546 Q2W (N=30) | 270 mg LY2541546 Q12W + Placebo (N=25) | Placebo Q2W (N=37)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Spinal cord ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 180 mg LY2541546 Q4W + Placebo (N=31) | 180 mg LY2541546 Q2W (N=30) | 270 mg LY2541546 Q2W (N=30) | 270 mg LY2541546 Q12W + Placebo (N=25) | Placebo Q2W (N=37)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 3 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (6) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 5 (5) | 3 (3) | 1 (1) | 2 (4)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Injection site bruising (General disorders) | 1 (4) | 3 (9) | 2 (7) | 6 (11) | 3 (3)
Injection site erythema (General disorders) | 3 (3) | 3 (5) | 2 (3) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Injection site induration (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 4 (7) | 5 (8) | 1 (2) | 1 (1) | 1 (1)
Injection site pruritus (General disorders) | 2 (2) | 5 (7) | 4 (5) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 6 (11) | 3 (5) | 5 (15) | 2 (3) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Asymptomatic bacteriuria (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (4) | 1 (1) | 2 (2) | 1 (2) | 2 (2)
Cystitis (Infections and infestations) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 2 (3)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 16 (20) | 8 (11) | 11 (19) | 7 (8) | 12 (16)
Oral herpes (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Pharyngitis (Infections and infestations) | 1 (1) | 3 (4) | 3 (3) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Respiratory tract infection viral (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 1 (3) | 2 (2) | 0 (0) | 5 (6)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Blood 1,25-dihydroxycholecalciferol increased (Investigations) | 6 (6) | 4 (5) | 4 (4) | 2 (2) | 5 (5)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urine calcium decreased (Investigations) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Urine phosphorus decreased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (5) | 2 (2) | 2 (2) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (4) | 2 (2) | 2 (2) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 3 (6) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (5)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (6) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (3) | 1 (1) | 2 (3) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 2 (2) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days